CLINICAL TRIAL: NCT04965415
Title: Small+Safe+Well: A Longitudinal Study of TWH in Small Business
Acronym: SSWell
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado School of Public Health (Other)
Collaborators: National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lee Newman, Distinguished professor, Colorado School of Public Health
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: U19OH011227 (NIH)
Record Dates: First submitted 2021-03-19; First posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Life Style

STUDY DESIGN:
Intervention Model Description: Businesses are randomly assigned to one of two arms, and the intervention is evaluated using a stepped wedge design. In the active comparator arm, businesses participate in an existing organizational-level intervention called Health Links in the first year of the study. Businesses randomly assigned to the experimental arm in the first year receive the TWH leadership program, in addition to Health Links. Businesses in the active comparator arm eventually receive the experimental intervention in the second year of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lagged (Active Comparator): Businesses in the lagged arm participated in Health Links for one year from their baseline assessment to their first follow-up assessment one year later. They were eligible to participate in the Leadership Training after both assessments were completed.
  Interventions: Behavioral: Health Links
- Early (Experimental): Businesses in this arm participated in Health Links + Leadership Training for one year from their baseline assessment to their first follow-up assessment one year later.
  Interventions: Behavioral: Health Links + Leadership Training

INTERVENTIONS:
Behavioral: Health Links + Leadership Training — Help businesses undergo transactional (i.e., business management practices) and transformational (i.e., business leadership and culture) change. Transactional change component: Health Links is an existing community-based intervention that seeks to help businesses - especially small and medium-sized businesses - incorporate Total Worker Health (TWH) programming into their business practices through assessment, advising, and certification. There is evidence that this consultation intervention is effective at helping businesses develop and implement policies and programs.Transformational change component: The experimental arm includes TWH leadership training for small business owners and other senior leaders. This is a three-month training that includes assessments, in-person training, and virtual training transfer activities. The goal is to help the leader understand their organization's current approach to TWH, identify areas for improvement, and to take action.
  Arms: Early
Behavioral: Health Links — Health Links is an existing community-based intervention that seeks to help businesses - especially small and medium-sized businesses - create a culture of both safety and health. Health Links does this by helping businesses incorporate Total Worker Health (TWH) programming into their business practices through assessment, advising, and certification. There is evidence that this consultation intervention is effective at helping businesses develop and implement policies and programs.
  Arms: Lagged

SUMMARY:
Workers in small businesses bear a disproportionate burden of occupational fatalities, illnesses, and injuries. The investigators conducted an intervention research project to determine how an intervention at the organizational level modifies business Total Worker Health (TWH) practices, safety climate, and health climate. In turn, the investigators aimed to determine whether organizational TWH adoption impacts individual workers' lifestyle health outcomes. In addition, the investigators also evaluated the use of the RE-AIM public health impact evaluation framework in the small business setting, with the intention of improving generalizability, maintenance, and dissemination of interventions and of guiding future TWH intervention design for both research and practice. The investigators conducted a lagged randomized controlled trial (L-RCT) to determine how different doses of an organizational-level TWH intervention (Health Links vs. Health Links + TWH Leadership Training) resulted in improvement and maintenance of TWH programming and organizational climates for safety and health, in small enterprises, over 36 months. The investigators also evaluated whether it resulted in improvements in workforce lifestyle health risks. In the short and mid-term, the goals and outputs of this project is a greater understanding of the theoretical underpinnings of TWH interventions and a model to test the implementation of the TWH interventions as well as an improvement the ability of TWH researchers and practitioners to apply this knowledge to TWH intervention design, implementation and evaluation to ensure generalizability. The long-term goal of this project is to impact worker safety, health and well-being through the continued use of these principles in small businesses.

ELIGIBILITY:
Inclusion Criteria:

* Colorado small business with less than 500 employees

Exclusion Criteria:

* Business does not operate in Colorado or has more than 500 employees

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2175 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Business Total Worker Health Policies and Programs | up to four years
  Total score, out of 100, on an assessment that measures the quantity of policies and programs that the business develops and implements to protect and promote their employees' health and safety.
Health Climate | up to four years
  Health climate (1-5 Likert scale, Strongly disagree to strongly agree) measures employee perceptions of whether their organization is committed to their health and well-being.
  Zweber, Z. M., Henning, R. A., & Magley, V. J. (2016). A practical scale for Multi-Faceted Organizational Health Climate Assessment. Journal of Occupational Health Psychology, 21(2), 250-259.
Safety Climate | up to four years
  Safety climate (1-5 Likert scale, Strongly disagree to strongly agree) measures employee perceptions of whether their organization is committed to their safety.
  Lee, J., Huang, Y.-H., Robertson, M. M., Murphy, L. A., Garabet, A., & Chang, W.-R. (2014). External validity of a generic safety climate scale for lone workers across different industries and companies. Accident Analysis & Prevention, 63, 138-145.
Overall health | up to four years
  A self-reported measure of overall health asks the respondent to rate their overall health (1-5 Likert scale, Poor to excellent).
  Schwatka, NV, Atherly, A, Dally, MJ, Fang, H, vS Brockbank, C, Tenney, L, Goetzel, RZ, Jinnett, K, Witter, R, Reynolds, S, McMillen, J, Newman, L. (2017). Health risk factors as predictors of workers' compensation claim occurrence and cost. Occupational and Environmental Medicine. 74(1): 14-23.
Well-being | up to four years
  A self-reported measure of well-being asks the respondent to rate their well-being related to mood (1-5 Likert scale, Poor to excellent).
  Staehr Johansen, K. (1998). The use of well-being measures in primary health care - the DepCare project. In World Health Organization, Regional Office for Europe: Well-Being Measures in Primary Health Care - The DepCare Project. Geneva, World Healthcare Organization.
Stress | up to four years
  A self-reported measure of stress asks the respondent to rate their level of stress related to work, home, and finances (1-5 Likert scale, Never to always).
  Schwatka, NV, Atherly, A, Dally, MJ, Fang, H, vS Brockbank, C, Tenney, L, Goetzel, RZ, Jinnett, K, Witter, R, Reynolds, S, McMillen, J, Newman, L. (2017). Health risk factors as predictors of workers' compensation claim occurrence and cost. Occupational and Environmental Medicine. 74(1): 14-23.
Sleep | up to four years
  A self-reported measure of sleep asks the respondent about the number of hours of sleep they get in a day (<6 hours, 6-6.9 hours, 7-8 hours, and >8 hours).
  Schwatka, NV, Atherly, A, Dally, MJ, Fang, H, vS Brockbank, C, Tenney, L, Goetzel, RZ, Jinnett, K, Witter, R, Reynolds, S, McMillen, J, Newman, L. (2017). Health risk factors as predictors of workers' compensation claim occurrence and cost. Occupational and Environmental Medicine. 74(1): 14-23.
Exercise | up to four years
  A self-reported measure of exercise asks the respondent about the number of days they get moderate to vigorous physical activity for at least 30 minutes.
  Schwatka, NV, Atherly, A, Dally, MJ, Fang, H, vS Brockbank, C, Tenney, L, Goetzel, RZ, Jinnett, K, Witter, R, Reynolds, S, McMillen, J, Newman, L. (2017). Health risk factors as predictors of workers' compensation claim occurrence and cost. Occupational and Environmental Medicine. 74(1): 14-23.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Newman, MA MA, Principal Investigator — Colorado School of Public Health
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
All business assessments and employee survey data collected by the researchers will be made available in a timely manner upon written request.
Supporting Information: Study Protocol
Time Frame: The data is currently available and will be stored in the longer term for three years after the study concludes (2023), per federal regulations.
Access Criteria: Files with de-identified data will be transferred via electronic format using a secure electronic file transfer along with a statement of data use standards. Documentation of data use standards will be included. To protect our participants we will make the data and its associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. The data will be stored in the longer term for three years after the study concludes, per federal regulations.

REFERENCES:
- [Background] Schwatka NV, Tenney L, Dally MJ, Scott J, Brown CE, Weitzenkamp D, Shore E, Newman LS. Small business Total Worker Health: A conceptual and methodological approach to facilitating organizational change. Occup Health Sci. 2018 Mar;2(1):25-41. doi: 10.1007/s41542-018-0013-9. PMID 30740514
- See also: Study website — https://coloradosph.cuanschutz.edu/research-and-practice/centers-programs/chwe/research/sswell